CLINICAL TRIAL: NCT03773705
Title: Impact of Nasoseptal Flap Harvest Technique on Olfaction Following Endoscopic Transsphenoidal Pituitary Surgery: A Single-blinded Randomized Controlled Trial
Brief Title: Impact of Nasoseptal Flap Harvest Technique on Olfaction Following Endoscopic Transsphenoidal Pituitary Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Unity Health Toronto (Other)
Responsible Party: Principal Investigator, John Lee, Head, Division of Rhinology, Principal Investigator, Unity Health Toronto
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 17-301
Record Dates: First submitted 2018-08-19; First posted 2018-12-12 (Actual); Last update posted 2019-03-15 (Actual); Status verified 2019-03

CONDITIONS: Pituitary Tumor; Surgery; Olfactory Nerve Injuries
MeSH Terms: conditions — Pituitary Neoplasms; Olfactory Nerve Injuries

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Electrocautery group (Active Comparator): Electrocautery used to raise pediclued nasoseptal flaps to repair skull based defects following endoscopic transphenoidal surgery.
  Interventions: Procedure: Electrocautery versus scalpel
- Scalpel group (Active Comparator): Scalpel used to raise pediclued nasoseptal flaps to repair skull based defects following endoscopic transphenoidal surgery.
  Interventions: Procedure: Electrocautery versus scalpel

INTERVENTIONS:
Procedure: Electrocautery versus scalpel — Electrocautery versus scalpel in the elevation of nasoseptal flaps following endoscopic transsphenoidal pituitary surgery

SUMMARY:
Pituitary tumours have an estimated prevalence of 20% in the general population and the number of clinically relevant pituitary adenomas is increasing with time. When symptomatic, the standard of care required for pituitary adenomas is resection through an endoscopic transsphenoidal approach. There is however significant olfactory dysfunction following endoscopic transsphenoidal pituitary surgery with approximately 23% of patients reporting some degree of worsening in their sense of smell in the postoperative period.

Pedicled nasoseptal flaps are used to repair skull base defects following resection of skull base tumours. The superior incision is placed in close proximity to olfactory mucosa. Currently, these flaps are raised either with the use of electrocautery or scalpel. The use of electrocautery in surgery has provided surgeons with greater hemostasis when compared to a scalpel. This is of utmost importance in many regions of the head & neck where highly vascularized tissue results in difficulties achieving adequate hemostasis and therefore limiting view of the surgical field. However, the use of electrocautery increases thermal damage to surrounding tissue and impairs wound healing when compared to a scalpel.

Although the transmission of thermal energy via electrocautery to adjacent mucosa containing olfactory epithelium may theoretically contribute to olfactory disturbances, no prospective randomized controlled trials have yet examined the impact of these two different techniques on postoperative olfactory function. The purpose of this research study is to determine the effects, if any, of electrocautery versus scalpel on olfaction in raising the nasoseptal flap for repairing skull base defects following transphenoidal surgery.

DETAILED DESCRIPTION:
Pedicled nasoseptal flaps are used to repair skull base defects following endoscopic transphenoidal surgery. The superior incision is placed in close proximity to olfactory mucosa. Currently, these flaps are raised either with the use of electrocautery or scalpel. While it is hypothesized that the olfactory mucosa is at greater risk of thermal injury with the use of electrocautery, no prospective multi-center studies have examined the impact of these two different techniques on postoperative olfactory function.

Patients will be recruited through the Otolaryngology-Head & Neck Surgery clinics. Based on previous studies in a North American population, a 10% change in UPSIT score was considered to be significant. With an alpha error set to 0.05, a beta of 0.8 and an effect size of 1 standard deviation, a sample size of 20 was calculated.

After obtaining consent for enrolment into the study, each patient will undergo either: (1) electrocautery or (2) scalpel in the elevation of nasoseptal flaps based on primary surgeon preference. The University of Pennsylvania Smell Identification Test (UPSIT) will be used for baseline testing of olfactory function in all enrolled patients. Postoperatively, all enrolled patients will be seen in follow-up at 1, 3 and 6 months' time, at which point the UPSIT will be administered for testing of postoperative olfactory function.

The Wilcoxon signed-rank test will be used to determine differences between UPSIT scores pre- and postoperatively. Results of p<0.05 will be considered statistically significant. Linear regression will be used to examine relationships between UPSIT scores and other variables collected (e.g., demographic data, size/type of pituitary tumour, length of nasoseptal flap).

Given that approximately 23% of all patients who undergo endoscopic transphenoidal surgery note some degree of worsening in their sense of smell following surgery, a prospective multi-center study comparing the two techniques would provide impetus to pursue one strategy over another in order to maintain an important sense, olfaction. Through optimizing preservation of olfactory mucosa during endoscopic skull base surgeries, patients' likelihood of not detecting environmental hazards (e.g., smoke, gas, other poisonous materials) will be reduced and, equally as important, their quality of life would be improved.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (age ≥18 years)
* Patients with tumours of the pituitary gland electively scheduled for endoscopic transsphenoidal surgery with nasoseptal flap coverage

Exclusion Criteria:

* Documented evidence of sinonasal disease on either nasal endoscopy or radiography
* Patients with a clinical history of asthma and/or sinonasal disease
* Previous sinus surgery
* Previous skull base surgery
* History of pre-existing hyposmia or anosmia
* Use of medication(s) known to alter sense of smell at time of test
* UPSIT scores <5 indicating a functional component to alteration in olfaction
* Development of postoperative cerebrospinal fluid leak necessitating re-entry into the operative field containing the nasoseptal flap

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2019-02-25 (Actual); Primary Completion 2019-10-31 (Estimated); Study Completion 2019-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in University of Pennsylvania Smell Identification Test (UPSIT) | Initial visit and at 1, 3 and 6-month follow-up visits
  Standardized and validated test of olfaction, which uses microencapsulated odorants released by scratching test booklets. Participants are asked to fill out forced choice multiple alternative questionnaires regarding each odorant. Minimum total score 0, maximum total score 40. Higher scores represent a better outcome.
Change in Sniffin' Sticks | Initial visit and at 1, 3 and 6-month follow-up visits
  Validated 16-item odor identification test. Minimum total score 0, maximum total score 16. Higher scores represent better outcome.
Change in Sino-Nasal Outcome Test-22 (SNOT-22) | Initial visit and at 1, 3 and 6-month follow-up visits
  Disease-specific, quality-of-life related measure of sinonasal function. Test consists of 22 symptoms requiring responders to rate severity on a 5-point Likert scale 0-5. Minimum score 0, maximum score 110. Higher scores correlate with greater rhinosinusitus-related health burden.
Change in Skull Base Inventory (SBI) | Initial visit and at 1, 3 and 6-month follow-up visits
  Multidimensional, disease-specific instrument designed to measure quality of life of patients who undergo surgical treatment for anterior or central skull base pathologies. It covers several disease-specific domains including cognitive, endocrine, nasal, neurologic, visual, and other general areas.Each item is weighted equally in each domain score. Each domain is weighted equally in the overall score. Domain scores are calculated by taking the total score (sum of all items) in that domain divided by the maximum possible score for that domain multiplied by 100. The minimum score for each domain is 0 and the maximum is 100. The minimum score for the questionnaire is 0 and the maximum is 100. Higher score indicates better outcomes.
Change in Pre-Op and Post-Op Endoscopy Scores | Initial visit and at 1, 3 and 6-month follow-up visits
  Used to quantify the pathological states of the nose and paranasal sinuses. Calculated on left and right side out, minimum 0, maximum 14. Higher scores indicate objectively worse sinonasal inflammation.

CONTACTS AND LOCATIONS:
Overall Officials: John Lee, MD, Principal Investigator — Unity Health Toronto
Locations (1):
- St. Michael's Hospital, Toronto, Ontario, Canada